CLINICAL TRIAL: NCT01248143
Title: Molecular and Clinical Effects of Green Tea and Fermented Papaya Preparation on Diabetes and Cardiovascular Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Touro College and University System (Other)
Collaborators: University of Mauritius (Other); Mauritius Cardiac Center (Unknown); Mauritius Ministry of Health and Quality of Life (Unknown); Osato Research Institute (Other); Societe Uniniere de Bois Cheri (Unknown); Mauritius Research Council (Other); University of Vienna (Other)
Responsible Party: Principal Investigator, Dr Okezie I Aruoma, Professor of Pharmaceutical and Biomedical Sciences, The Touro College and University System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPP and TEA IN DIABETES
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Assess the Effect of Green Tea on Diabetes; Assess the Effect of Fermented Papaya Pretration on Diabetes; Effects of Green Tea and FPP on C-reactive Proteins; Effects of Green Tea and FPP of Lipid Profiles in Diabetes; Effect of Green Tea and FPP on Atheroma Formation
Keywords: Green Tea; Fermented papaya preparation; Diabetes; Cardiovascular diseases; Atherosclerotic plaques; Glucose; Dietary supplements and functional foods
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Plaque, Atherosclerotic | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green tea (Experimental)
  Interventions: Dietary Supplement: Green tea
- FPP (Experimental)
  Interventions: Dietary Supplement: FPP

INTERVENTIONS:
Dietary Supplement: Green tea — 9 gram per day
  Arms: Green tea
Dietary Supplement: FPP — 2 sachets twice daily
  Arms: FPP

SUMMARY:
Type 2 diabetes is common in ethnic and, minority groups in developing and developed countries such as Africans, African Americans, Asians, Native Americans, Hispano-Latinos and Alaskan indians. A randomized controlled study to assess the efficacy of fermented papaya preparation and green tea infusates in latent diabetes (individuals newly diagnosed as diabetics) is proposed. Glycation products from excess glucose autooxidation can chemically modify DNA causing mutations and cause complex DNA rearrangements. Advanced glycation end-products which play a role as proinflammatory mediators in gestational diabetes can accelerate vascular occlusion by quenching the vasodilating agent nitric oxide. Interaction with high-affinity receptors located on monocytes and macrophages can enhance the production of free radicals and reactive oxygen/nitrogen species, the secretion of tumor necrosis factor-α, interleukin-1 and insulin-like growth factor I which can proliferate endothelial, mesangial and smooth muscle cells and hence contribute significantly to the pathogenesis of cardiovascular complications. The clinical markers include C-reactive proteins (inflammation indicators), protein C (markers of reno vascular injury), uric acid, natriuretic peptides, and the integrity of isolated adipocytes, glucose levels, lipid indices (triglycerides, total cholesterol, VLDL, HDL and LDL). Given that decreased functional activity of activated protein C affects the permeability of the glomerular capillary wall and enhances apoptosis of glomerular endothelial cells and adipodocytes, this has relevance to the pathophysiology of diabetic nephropathy. A second phase of the study is expected to commence after the first 16 weeks in order to assess the ability of the dietary factors to modulate atheroma formation and the integrity of drug therapy (upon commencement of treatment)on the prognosis of diabetes. This will be expected to last up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

Individuals at risk of diabetes 35-65 years of age male or female

Exclusion Criteria:

* Smokers or those who have stopped smoking 6 months before the study
* Daily alcoholic intake exceeding 4 standard drinks
* Post menopausal women currently under hormone replacement treatment
* Hypertension (>140/90 mm Hg)
* individuals outside the age range 35-60

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Assess the effects of green tea and FPP on the levels of C-reactive proteins | 3 months
  The pathophysiology of atherosclerosis and other cardiovascular events have associated inflammatory processes. The levels of plasma high-sensitivity (hs) C-Reactive Protein, an acute phase reactant produced in the liver, known to rise in inflammatory reactions are widely suggested to be a predictor of coronary events; and increased uric acid levels (hyperuricemia) are considered to be a risk factor in many clinical conditions including hypertension, cardiovascular events, diabetes mellitus, stroke, and metabolic syndrome.

SECONDARY OUTCOMES:
Assess the effect of green tea and fermented papaya preparation on development of atheroma and drug therapy outcomes | 3 years
  Carotid artery angioplasty and stenting has been proposed as an alternative therapy for patients requiring treatment of carotid artery stenosis as opposed to the "gold standard" surgical intervention, carotid endarterectomy. The second phase of the study will investigate the possible role of green tea and fermented papaya preparation in modulating the risk of stroke by assessing the extent of atheroma using both echocardiography and CT angiography. Patients will be on medication and the therapeutic outcome will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Okezie I Aruoma, PhD DSc, Principal Investigator — Touro College of Pharmacy
Locations (3):
- Touro College of Pharmacy, New York, New York, United States
- University of Vienna, Vienna, Austria
- University of Mauritius, Réduit, Mauritius

REFERENCES:
- [Background] Bahorun T, Luximon-Ramma A, Gunness TK, Sookar D, Bhoyroo S, Jugessur R, Reebye D, Googoolye K, Crozier A, Aruoma OI. Black tea reduces uric acid and C-reactive protein levels in humans susceptible to cardiovascular diseases. Toxicology. 2010 Nov 28;278(1):68-74. doi: 10.1016/j.tox.2009.11.024. Epub 2009 Dec 4. PMID 19963031
- [Result] Bahorun T, Luximon-Ramma A, Neergheen-Bhujun VS, Gunness TK, Googoolye K, Auger C, Crozier A, Aruoma OI. The effect of black tea on risk factors of cardiovascular disease in a normal population. Prev Med. 2012 May;54 Suppl:S98-102. doi: 10.1016/j.ypmed.2011.12.009. Epub 2011 Dec 16. PMID 22198621
- [Result] Somanah J, Aruoma OI, Gunness TK, Kowelssur S, Dambala V, Murad F, Googoolye K, Daus D, Indelicato J, Bourdon E, Bahorun T. Effects of a short term supplementation of a fermented papaya preparation on biomarkers of diabetes mellitus in a randomized Mauritian population. Prev Med. 2012 May;54 Suppl:S90-7. doi: 10.1016/j.ypmed.2012.01.014. Epub 2012 Feb 11. PMID 22330753
- [Result] Toolsee NA, Aruoma OI, Gunness TK, Kowlessur S, Dambala V, Murad F, Googoolye K, Daus D, Indelicato J, Rondeau P, Bourdon E, Bahorun T. Effectiveness of green tea in a randomized human cohort: relevance to diabetes and its complications. Biomed Res Int. 2013;2013:412379. doi: 10.1155/2013/412379. Epub 2013 Sep 12. PMID 24102055
- [Result] Somanah J, Bourdon E, Rondeau P, Bahorun T, Aruoma OI. Relationship between fermented papaya preparation supplementation, erythrocyte integrity and antioxidant status in pre-diabetics. Food Chem Toxicol. 2014 Mar;65:12-7. doi: 10.1016/j.fct.2013.11.050. Epub 2013 Dec 5. PMID 24316314
- [Result] Aruoma OI, Somanah J, Bourdon E, Rondeau P, Bahorun T. Diabetes as a risk factor to cancer: functional role of fermented papaya preparation as phytonutraceutical adjunct in the treatment of diabetes and cancer. Mutat Res. 2014 Oct;768:60-8. doi: 10.1016/j.mrfmmm.2014.04.007. Epub 2014 Apr 24. PMID 24769427